CLINICAL TRIAL: NCT03296917
Title: A Phase II, Double-Blinded, Randomised, Controlled Study to Examine the Prophylactic Efficacy, Safety and Tolerability of PrEP-001 in Asthmatic Subjects Subsequently Challenged With Human Rhinovirus (HRV-16)
Brief Title: Study Examining PrEP-001 in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hvivo (Industry)
Collaborators: Prep Biopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PrEP-CS-002
Record Dates: First submitted 2017-06-13; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — G004 compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMP - PrEP-001 (Experimental): In Viral Challenge arm cohort:
  A nasal dose of 6400 μg PrEP-001 equally divided over both nostrils on 2 consecutive days (Day -2 and Day -1).
  In the Safety arm's first dose cohort:
  A nasal dose of 6400 μg PrEP-001 equally divided over both nostrils on 2 consecutive days (Day -2 and Day -1).
  Then assuming no significant safety issues with the lower dose (as determined by blinded review by the DSMB team), the Safety arm's second dose cohort will consist of:
  A nasal dose of 12800 μg PrEP-001 equally divided over both nostrils on 2 consecutive days (Day -2 and Day -1)
  Interventions: Drug: PrEP-001
- Placebo - G-004 (Placebo Comparator): In the Viral Challenge arm and each Safety Arm cohort:
  A nasal dose of placebo equally divided over both nostrils on 2 consecutive days (Day -2 and Day -1).
  Interventions: Drug: G-004

INTERVENTIONS:
Drug: PrEP-001 — A spray dried powder for intranasal administration formulated from an aqueous mixture of pre-gelatinized waxy maize starch and the drug substance delivered using a single dose nasal powder device.
  Arms: IMP - PrEP-001
Drug: G-004 — A spray dried pre-gelatinized waxy maize starch powder (G-001) in the single dose nasal powder device
  Arms: Placebo - G-004

SUMMARY:
Phase 2 study, to examine the prophylactic efficacy, safety and tolerability of PrEP-001 in asthmatics who have been infected with the human rhinovirus (HRV16) after receiving two doses of the study drug/placebo.

DETAILED DESCRIPTION:
Screening took place up to 90 days before quarantine, where volunteers were asked to complete an informed consent and undergo scheduled screening assessments to determine their eligibility.

Eligible volunteers were invited to test and record their respiratory symptoms and peak expiratory flow (PEF), medications and any adverse events in diary cards from Day -14 to Day -5.

They attended Quarantine on Day -4/-3, received the study drug/placebo intra nasally on Day -2 and Day -1 and subsequently challenged with HRV16 on Day 0. Randomisation to receive study drug/placebo was 1:1.

Volunteers remained in the quarantine unit for 8 days after inoculation.

PEF self-testing continued from Day 9 to Day 28.

On Day 20 (±3 days) and Day 28 (±5 days), volunteers attended follow up visits where they were assessed by a study physician for well-being, on-going symptoms and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years on the day of first dosing with IMP.
* Physician diagnosed asthma for at least 6 months prior to Screening and using treatment equivalent up to and including Global Initiative for Asthma (GINA) Stage 3.
* In good health with no history of major medical conditions (other than asthma) that will interfere with subject safety, as defined by medical history, physical examination, and routine laboratory tests as determined by the Investigator at a screening evaluation.

Exclusion Criteria:

* Any ex-smoker or smoker with a history of more than 10 pack-years.
* History of life-threatening asthma, Diagnosis of COPD as defined by the current Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2014 guidelines.
* Any history or evidence of any clinically significant medical and psychiatric conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: The Area Under the Curve (AUC) of total symptom score post viral challenge. | Day -14 to Day 28
  AUC of total symptom scores (upper respiratory tract (URT), lower respiratory tract (LRT) and systemic viral symptoms (SVS)). Total symptom scores (from the symptom diary card) used to calculate the AUC. The primary endpoint is only being derived from the Viral Challenge arm.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint: Symptom Scores: Area Under the Curve (AUC) | Day -4 to Day 28
  AUC of individual symptom scores (upper respiratory tract (URT), lower respiratory tract (LRT) and systemic viral symptoms (SVS)). A total symptom score is derived for each subject, separately for each assessment (symptom diary card) on each day.
Secondary Efficacy Endpoint: Symptom Scores: Duration of symptoms | Day -4 to Day 28
  Time (days).
Secondary Efficacy Endpoint: Symptom Scores: Peak symptoms score | Day -4 to Day 28
  Numerical sum of all individual composite symptoms.
Secondary Efficacy Endpoint: Symptom Scores: Time to peak symptoms | Day -4 to Day 28
  Time (days).
Secondary Efficacy Endpoint: Symptom Scores: Time to resolution from peak symptoms | Day -4 to Day 28
  Time (days).
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: viral shedding | Day -4 to Day 28
  Number of subjects with viral shedding.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: incidence of laboratory-confirmed Influenza illness | Day -4 to Day 28
  The number of subjects with laboratory-confirmed influenza infection.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: laboratory confirmed Influenza A/Perth/16/2009 (H3N2) Virus infection | Day -4 to Day 28
  The number of subjects with laboratory-confirmed influenza A/Perth/16/2009 (H3N2) Virus infection.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: HRV-like-illness | Day -4 to Day 28
  The number of subjects with HRV-like illness.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: Sub-clinical infection | Day -4 to Day 28
  The number of subjects with Sub-clinical illness.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: Upper respiratory tract illness | Day -4 to Day 28
  The number of subjects with Upper respiratory tract illness.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: Lower respiratory tract illness | Day -4 to Day 28
  The number of subjects with Lower respiratory tract illness.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: Febrile illness | Day -4 to Day 28
  The number of subjects with Febrile illness.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: Systemic illness | Day -4 to Day 28
  The number of subjects with Systemic illness.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: Non-sick and uninfected | Day -4 to Day 28
  The number of subjects Non-sick and uninfected.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: Viral replication, as measured by tissue culture assay | Day -4 to Day 28
  The number of subjects with viral replication.
Secondary Efficacy Endpoint: Incidence(s) of illness and infection: Seroconversion | Day -4 to Day 28
  The number of subjects with seroconversion.
Secondary Efficacy Endpoint: Viral Load Parameters: Area under the curve (AUC) of viral load, as measured by nasopharyngeal swab RT-qPCR | Day -4 to Day 28
  Viral load data supplied in Log10 Copies/mL. These values used to calculate the Area Under the Curve (AUC) for each subject.
Secondary Efficacy Endpoint: Duration of virus shedding, as measured by nasal wash RT-qPCR | Day -4 to Day 28
  Time (days).
Secondary Efficacy Endpoint: Peak virus shedding, as measured by nasal wash RT-qPCR | Day -4 to Day 28
  The highest observed RT-qPCR viral load value.
Secondary Efficacy Endpoint: Viral Load Parameters: Time to peak viral shedding, as measured by nasal wash RT-qPCR | Day -4 to Day 28
  Time (days).
Secondary Efficacy Endpoint: Time to resolution from peak viral shedding, as measured by nasal wash RT-qPCR. | Day -4 to Day 28
  Time (days).
Secondary Efficacy Endpoint: Area under the curve (AUC) of viral load, as measured by nasal wash TCID50. | Day -4 to Day 28
  Tissue culture viral load data supplied in log10 TCID50/mL. These values used to calculate the Area Under the Curve (AUC) for each subject.
Secondary Efficacy Endpoint: Duration of virus shedding, as measured by nasal wash TCID50. | Day -4 to Day 28
  Time (days).
Secondary Efficacy Endpoint: Peak virus shedding, as measured by nasal wash TCID50. | Day -4 to Day 28
  The highest observed RT-qPCR viral load value.
Secondary Efficacy Endpoint: Time to peak viral shedding, as measured by nasal wash TCID50. | Day -4 to Day 28
  Time (days).
Secondary Efficacy Endpoint: Total weight of nasal discharge produced post Viral Challenge to Quarantine discharge. | Day -4 to Day 28
  Weight (grams).
Secondary Efficacy Endpoint: Change in lung function compared to pre-Challenge. | Day -4 to Day 28
  Peak Expiratory Flow (L/min) and FEV1 (L)
Secondary Efficacy Endpoint: Change in Asthma Control Questionnaire (ACQ) score compared to pre-Challenge. | Day -4 to Day 28
  ACQ score.
Secondary Efficacy Endpoint: Change in Fractional exhaled nitric oxide (FeNO) compared to pre-Challenge. | Day -4 to Day 28
  FeNO (ppb).

OTHER OUTCOMES:
Exploratory Efficacy Analysis: Proportion (on any occasion) of subjects with Grade 2 or worse symptoms at any day post-Viral Challenge. | Day -14 to Day 28
  Number of subjects with Grade 2 or higher symptoms at any day post-Viral Challenge.
Exploratory Efficacy Analysis: Proportion of subjects with Grade 2 or worse symptoms at each day post-Viral Challenge. | Day -4 to Day 28
  Number of subjects with symptoms at Grade 2 or higher, at each day post-Viral Challenge.
Exploratory Efficacy Analysis: Duration of Grade 2 or worse symptoms (post-Viral Challenge). | Day -4 to Day 28
  Time (days).
Exploratory Efficacy Analysis: Proportion of subjects with any clinical symptoms (i.e., with Grade ≥ 1) (post-Viral Challenge). | Day -4 to Day 28
  The proportion of subjects with symptoms grade 1 or higher.
Exploratory Efficacy Analysis: Proportion of subjects with Grade ≥1 symptom score for upper respiratory tract (URT) symptoms (post-Viral Challenge). | Day -4 to Day 28
  The proportion of subjects with upper respiratory tract symptoms.
Exploratory Efficacy Analysis: Proportion of subjects with Grade ≥1 symptom score for lower respiratory tract (LRT) symptoms (post-Viral Challenge). | Day -4 to Day 28
  The proportion of subjects with lower respiratory tract symptoms.
Exploratory Efficacy Analysis: Proportion of subjects with Grade ≥1 symptom score for systemic symptoms (post-Viral Challenge). | Day -4 to Day 28
  The proportion of subjects with systemic symptoms.
Exploratory Efficacy Analysis: Time to peak for each reported and any symptoms (post-Viral Challenge). | Day -4 to Day 28
  Time (days).
Exploratory Efficacy Analysis: Proportion of subjects with pyrexia. | Day -4 to Day 28
  The proportion of subjects with pyrexia.
Exploratory Efficacy Analysis: Duration of pyrexia. | Day -4 to Day 28
  Time (hours).
Exploratory Efficacy Analysis: Tympanic temperature. | Day -4 to Day 28
  Changes in tympanic temperature over time (post Viral Challenge) (degrees Celcius)
Exploratory Efficacy Analysis: Area under the curve (AUC) of symptom scores using the 13-item symptom diary card (total, URT, LRT and SVS), Day 1 (assessment 1) to Day 8. | Day -4 to Day 28
  AUC of individual symptom scores.
Exploratory Efficacy Analysis: Proportion of subjects with Lab-confirmed Clinical Symptoms of URTI. | Day -4 to Day 28
  The number of subjects with lab-confirmed clinical symptoms of URTI.
Exploratory Efficacy Analysis: Proportion of subjects with Lab-confirmed Clinical Symptoms of LRTI. | Day -4 to Day 28
  The number of subjects with lab-confirmed clinical symptoms of LRTI.
Exploratory Efficacy Analysis: Proportion of subjects with Lab-confirmed Clinical Symptoms of Systemic Illness (SI). | Day -4 to Day 28
  The number of subjects with lab-confirmed clinical symptoms of SI.
Exploratory Efficacy Analysis: Overall total symptom score, Day 1 (assessment 1) to Day 8, using the 10-item symptom diary card. | Day -4 to Day 28
  Total symptom score.
Exploratory Efficacy Analysis: Overall symptom scores (URT, LRT SVS), Day 1 (assessment 1) to Day 8, using the 10-item symptom diary card. | Day -4 to Day 28
  Total symptom score.
Safety endpoint: Treatment-emergent Adverse Events (TEAE). | Day -4 to Day 28
  Incidence of treatment-emergent AEs (TEAE), overall, and by severity and causality (analysed descriptively).
Safety endpoint: Clinical laboratory parameters. | Day -4 to Day 28
  Absolute values and change from baseline in routine clinical laboratory parameters by timepoint (analysed descriptively). Includes haematology, biochemistry, coagulation, cardiac enzymes, thyroid function tests and urinalysis parameters.
Safety endpoint: Vital signs. | Day -4 to Day 28
  Absolute values and change from baseline in vital signs parameters by timepoint (analysed descriptively); systolic blood pressure (SBP) (mmHg), diastolic blood pressure (DBP) (mmHg), respiratory rate (RR) (breaths per minute), heart rate (HR) (beats per minute) and SpO2 (%).
Safety endpoint: Physical Examination. | Day -4 to Day 28
  Physical examination findings (analysed descriptively).
Safety endpoint: Spirometry. | Day -4 to Day 28
  Absolute and changes from baseline for FEV1 [absolute] (L), FEV1 [% predicted] (%), FVC [absolute] (L), FVC [% predicted] (%), FEV1/FVC ratio [absolute], FEV1/FVC ratio [% predicted] (%), maximum mid expiratory flow (MMEF) [absolute] (L/sec) and MMEF [% predicted]). The lung function parameter Peak Expiratory Flow [L/min] will also be summarised (analysed descriptively).
Safety endpoint: ECGs. | Day -4 to Day 28
  12-lead electrocardiogram (ECG) findings (analysed descriptively).
Safety endpoint: Asthma Exacerbations (Number) | Day -4 to Day 28
  Number and percentage of subjects experiencing any asthma exacerbations.
Safety endpoint: Duration of each asthma exacerbation | Day -4 to Day 28
  Time (days)
Safety endpoint: Time to first asthma exacerbation | Day -4 to Day 28
  Time (days)
Safety endpoint: Subjects requiring treatment for asthma exacerbation | Day -4 to Day 28
  Number of subjects requiring oral or parenteral steroids as treatment for their exacerbation.
Safety endpoint: Subjects requiring hospitalisation for asthma exacerbation | Day -4 to Day 28
  Number of subjects requiring hospitalisation for their exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: John Efthimiou, Study Chair — Sponsor's Representative